CLINICAL TRIAL: NCT00738959
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD0328 in Healthy Young Japanese and Caucasian Male Volunteers After Oral Single and Multiple Ascending Doses
Brief Title: Safety, Tolerability & PK of AZD0328 in Caucasian & Japanese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Didier Meulien, MD, Medical Science Director, Emerging AD & Cognition, AstraZeneca R&D, Södertälje, Sweden
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: D0190C00008; EUdract NO 2008-001723-56
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Healthy Volunteers
Keywords: AZD0328; Japanese; Caucasian; pharmacokinetics; safety; tolerability
MeSH Terms: interventions — spiro(1-azabicyclo(2.2.2)octane-3,2'(3H)-furo(2,3-b)pyridine)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD0328

INTERVENTIONS:
Drug: AZD0328 — Oral solution A single dose Day 1 followed by once daily doses on Day 3-7

SUMMARY:
This study will be performed to evaluate the safety, tolerability and pharmacokinetics of single and multiple doses of AZD0328 when administered to Japanese and Caucasian healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* first generation Japanese (both parents and grandparents are Japanese, the subject is born in Japan and left Japan less than 10 years ago) or Caucasian subjects.
* Clinically normal physical findings, laboratory values, vital signs and resting ECG as judged by the investigator.

Exclusion Criteria:

* History of clinically significant cardio- or cerebrovascular, pulmonary, renal, hepatic, neurological, mental or gastrointestinal disorder or any other major disorder that may interfere with the study.
* Participation in another study within 12 weeks before the first administration of the investigational product.
* Intake of any prescribed medicine or herbal remedies based on St John's Wort, except for occasional paracetamol and nasal adrenergic anticongestants, within 3 weeks before the first administration of the investigational product.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, paper ECGs and 12-lead continuous digital ECGs including QT/QTc interval measurements | During the whole treatment period

SECONDARY OUTCOMES:
PK variables | Several samples during the study days

CONTACTS AND LOCATIONS:
Overall Officials: Didier Meulien, MD, Study Director — AstraZeneca R&D Södertälje, Sweden; Ulrike Lorch, MD, Principal Investigator — Richmond Pharmacology Ltd St George's University of London Cranmer Terrace, TootingLondon SW17 ORE UK
Locations (1):
- Research Site, London, United Kingdom